CLINICAL TRIAL: NCT07093320
Title: Immediate Vascular and Soft Tissue Reconstruction After Sarcoma Resection Involving Major Limb Vessels: Early and Midterm Outcomes From a Tertiary Center
Brief Title: Saving Limbs After Cancer: Blood Vessel and Soft Tissue Reconstruction Following Sarcoma Surgery in the Legs
Acronym: SARCOVASCPLAST
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Martin Lhuaire, Dr, European Georges Pompidou Hospital
Other Study IDs: SARCOVAPLAST; number IRB 00006477 (Other: Hôpitaux Universitaires Paris Nord Val de Seine AP-HP)
Record Dates: First submitted 2025-07-15; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma (STS)
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STS with major vessel involvement: STS with major vessel involvement
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aimed to evaluate whether immediate reconstruction of blood vessels and soft tissues can safely and effectively preserve limbs in patients undergoing surgery for sarcomas involving major arteries or veins in the arms or legs. The goal was to determine if this complex surgical approach helps avoid amputation, ensures good cancer control, and leads to acceptable complication rates and healing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patient presented with STS with major vessels involvement

Exclusion Criteria:

* All STS without major vessels involvement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary center (sarcoma reference center), teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
1- Limb salvage rate 2- Flap survival 3- Vascular patency | At 12 months postoperatively
  1. Limb salvage: Determined by clinical documentation of limb preservation without major amputation.
  2. Flap survival: Determined by clinical evaluation of flap viability
  3. Vascular patency: Determined by duplex ultrasonography or CT angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Martin LHUAIRE, MD, Msc, Principal Investigator — Service de Chirurgie Plastique, Reconstructrice et Esthétique, Hôpital Européen Georges Pompidou Paris, , France 75015; Laurent Lantieri, MD, Study Chair — Service de Chirurgie Plastique, Reconstructrice et Esthétique, Hôpital Européen Georges Pompidou Paris, , France 75015; David BIAU, MD, PhD, Study Director — Service de Chirurgie Orthopédique et oncoorthopédie, Hôpital Cochin, Paris, , France 75015
Locations (1):
- Service de Chirurgie Plastique, Reconstructrice et Esthétique, Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after publication of the data
Access Criteria: De-identified individual participant data (IPD) and supporting documentation will be made available by the Principal Investigator upon reasonable request from qualified researchers.
URL: https://www.aphp.fr